CLINICAL TRIAL: NCT04695834
Title: A Prospective, Multi-center, Randomized, Parallel-group Controlled Trial to Compare Conservative Versus Surgical Treatment of Foot Drop in Peroneal Nerve Entrapment.
Brief Title: Follow-up and Outcome of Operative Treatment With Decompressive Release Of The Peroneal Nerve
Acronym: FOOTDROP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Health Care Knowledge Centre (KCE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S62895; KCE19-1232 (Other Grant/Funding Number: KCE Belgium)
Record Dates: First submitted 2020-12-03; First posted 2021-01-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Peroneal Nerve Entrapment
Keywords: Peroneal nerve; Neurolysis; Conservative treatment; Randomised controlled trial; Foot drop
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Intervention Model Description: Prospective Multi-center Randomized Parallel-group
Who Masked: Outcomes Assessor
Masking Description: All participants will be asked to wear long trousers to cover a potential scar at the level of the knee.
  All patients will be asked to apply a bandage at the site of the operation (or the site of entrapment if there was no operation) Participants are not allowed to discuss their treatment with the outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (Active Comparator): Patients that are randomized to the conservative arm of the trial. These patients will not be operated until primary endpoint is reached.
  If necessary, cross-over can occur after primary endpoint is reached.
  Conservative treatment is considered standard of care.
  Interventions: Other: Maximal physiotherapy
- Surgical treatment (Active Comparator): Patients randomized to the surgical arm will be operated within 1 week after randomization (if possible within 2 days).
  Neurolysis is considered standard of care.
  Interventions: Procedure: Neurolysis peroneal nerve

INTERVENTIONS:
Procedure: Neurolysis peroneal nerve — The surgical approach for entrapment at the fibular head is usually through a curvilinear incision just distal to the fibular head. The subcutaneous tissue is bluntly dissected, and the common peroneal nerve is identified proximal to the peroneus longus muscle. The peroneal nerve is then released from the surrounding fibrous tissue and fascia. The nerve is decompressed distally as it dives under the peroneus longus muscle. The decompression at this site is essential. Certain authors state that an adequate decompression should extend beyond the bifurcation in the deep and superficial peroneal nerve and should involve cutting the intermuscular septa
  Arms: Surgical treatment
Other: Maximal physiotherapy — Mobilization of ankle and foot, stretching of the calf muscles (prevention of contractures) Tonification of the dorsiflexion- and eversion muscles of the ankle Proprioceptive training Gait rehabilitation Home exercise schedule
  Arms: Conservative treatment

SUMMARY:
The FOOT DROP trial is a prospective, multi-center, randomized controlled trial to assess if decompressive surgery for peroneal nerve entrapment is superior to maximal conservative treatment.

Patients with persisting foot drop due to peroneal nerve entrapment will be randomized to either surgery or conservative treatment if foot drop persists 10 +/- 4 weeks after onset of symptoms.

Patients will be evaluated through several questionnaires, evolution of muscle strength and several types of gait assessments. Primary endpoint is the difference in distance covered during the six minute walking test between baseline and 9 months after randomization.

DETAILED DESCRIPTION:
The Foot Drop Trial is the first prospective, randomised controlled trial to investigate the treatment of foot drop in peroneal nerve entrapment. Currently, the literature consists mostly of biased retrospective case series with the exception of some small (biased) prospective case series. No comparative trials have been conducted. The goal of the trial is to assess whether foot drop due to peroneal nerve entrapment recovers better 9 months after decompressive surgery compared to maximal conservative treatment.

Patients with persisting foot drop (MRC score ankle dorsiflexion ≤ 3) after 10 +/- 4 weeks after onset of symptoms will be randomised to either decompressive surgery within 1 week after randomisation or maximal conservative treatment focussing on physiotherapy and gait rehabilitation. Blinded outcome assessors will evaluate participants at study visits 10 days (surgical group), 6 weeks, 3 months, 6 months, 9 months (primary outcome) and 18 months (extended follow-up) after randomization.

Outcome assessors will conduct several assessments to evaluate gait improvement (6-minute walk test, 10-meter walk test, Stanmore questionnaire, functional ambulation categories, ability to walk barefoot, need for foot-ankle orthosis), muscle strength (MRC score for ankle dorsiflexion, ankle eversion, hallux extension) , quality of life (EQ-5D 5L) and cost-effectiveness of both treatment strategies (work productivity and activity impairment questionnaire (WPAI), return to work, percentage of invalidity). Electrodiagnostic follow-up will be registered at 3 months and 9 months after randomization.

The primary endpoint of the foot drop trial is the difference in distance covered in meters during the six-minute walk test (6MWD) between baseline and 9 months after randomization. Time to recovery, defined as the time necessary to cover the minimal age- and sex-specific normal 6MWD AND the time necessary for foot drop recovery to an MRC-score ≥ 4 for ankle dorsiflexion is the key secondary endpoint. No cross-over to surgery is allowed before primary endpoint is reached.

The study first succesfully piloted in 6 centers in Belgium and the Netherlands and is currently starting on a large scale in 20 centers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study must be obtained from the subject or proxy / legal representative prior to initiation of any study-mandated procedure
* EDX-documented peroneal nerve entrapment with persisting (10 ± 4 weeks) foot drop (MRC-score ≤ 3)
* Imaging (ultrasound/MRI) performed to exclude a compressive mass
* Age ≥ 18 years

Exclusion Criteria:

* Subjects with posttraumatic or iatrogenic peroneal nerve injury
* Subjects with peroneal neuropathy due to a compressive mass (e.g. cyst, tumour)
* Peroneal nerve entrapment at other sites than the fibular head
* Patients with mental or physical problems that incapacitate them to participate in a physiotherapy program
* Psychiatric illness
* Pregnancy
* Planned (e)migration within 1 year after randomization to another country
* Subjects with previous foot drop
* Permanently bedridden subjects
* Subjects with neurological or musculoskeletal history which could impact foot drop assessment and/or gait analysis (e.g. polyneuropathy, hereditary neuropathy with pressure palsies, critical illness polyneuropathy, previous stroke, ankle surgery, …).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in distance covered in meters during the six-minute walk test (6MWD) between baseline and 9 months after randomization. | 9 months
  Based on a literature analysis and patient feedback on the trial design, gait analysis and recovery of a normal gait pattern are crucial in the recovery of foot drop. In 90% of interviewed patients, success of treatment was related to improvement in gait. The distance covered during the six-minute walk test (6MWT) is validated and clinically used in gait analysis.
  6MWT: patients are instructed to walk as far as possible within six minutes (strokes of 30 meters of more).
  The minimal age- and sex-specific normal 6MWD is defined as 82% of the applied reference equations for prediction of the 6MWD. The reference value that will be used is 6MWDpred(m) = 868.8 - (ageyears x 2.99) - (gender x 74.7). The value for gender is 0 in male subjects and 1 in female subjects.

SECONDARY OUTCOMES:
Time to recovery | 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  KEY SECONDARY ENDPOINT Time to recovery is defined as: the time necessary to cover the minimal age- and sex-specific normal distance in meters during the 6-minute walking test (6MWT) AND the time necessary for foot drop recovery to an MRC-score ≥ 4 for ankle dorsiflexion.
  The MRC-score is a clinical assessment of muscle strength. MRC-ranges from 0 to 5 with zero indicating no movement at all and 5 indicating normal muscle strength.
  The minimal age- and sex-specific normal 6-minute walking distance (6MWD) is defined as 82% of the applied reference equations for prediction of the 6MWD. The reference value that will be used is 6MWDpred(m) = 868.8 - (ageyears x 2.99) - (gender x 74.7). The value for gender is 0 in male subjects and 1 in female subjects.
Ankle dorsiflexion strength as measured by the Medical Research Council score (MRC-score). | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization))
  Medical Research Council (MRC)-score as clinical assessment of muscle strength. MRC-score ranges from 0 to 5.
  0: no movement
  1. contraction of muscle, but no movement
  2. movement, but not against gravity
  3. movement against gravity, but not against resistance
  4. movement against resistance
  5. normal strength
Ankle dorsiflexion strength as measured by isometric dynamometry. | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization))
  Recovery of ankle dorsiflexion strength is essential in patients with foot drop. The use of dynamometry allows to document ankle dorsiflexion strength in an objective manner.
  Patients are asked to lay in supine position, with the knees extended. The test pad of the dynamometer is placed on the dorsal head of the first metatarsal bone. The patient is instructed to perform ankle dorsiflexion with maximal muscle strength. The best of three attempts is registered. Ankle dorsiflexion is measured and reported in both ankles (in kilograms). The ankle dorsiflexion strength ratio, defined as the ratio of ankle dorsiflexion strength in the affected ankle over ankle dorsiflexion strength in the healthy ankle will be calculated and reported
Complications and neurologic deficits: Motor changes as assessed by the Medical Research Council Score (MRC-score) for hallux extension | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization))
  Medical Research Council (MRC)-score as clinical assessment of muscle strength. MRC-score ranges from 0 to 5.
  0: no movement
  1. contraction of muscle, but no movement
  2. movement, but not against gravity
  3. movement against gravity, but not against resistance
  4. movement against resistance
  5. normal strength
Complications and neurologic deficits: Sensory changes | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization))
  In a large retrospective patient series on peroneal nerve decompression after weight loss, Broekx et al. (2018) examined the recovery of sensory deficits. Symptoms qualified as sensory included the presence of hypoesthesia and/or paresthesia. They used the following system to assess sensory symptoms:
  1. Complete recovery: the absence of any sensory symptoms
  2. Partial recovery: patients with a minimum of sensory symptoms
  3. No recovery: patients with no improvement
Gait assessment: Difference in distance covered in meters during the six-minute walk test | 6 weeks, 3 months, 6 months and 18 months (after randomization)
  The distance covered during the six-minute walk test (6MWT) is validated and clinically used in gait analysis.
  6MWT: patients are instructed to walk as far as possible within six minutes (strokes of 30 meters of more).
  The minimal age- and sex-specific normal 6MWD is defined as 82% of the applied reference equations for prediction of the 6MWD. The reference value that will be used is 6MWDpred(m) = 868.8 - (ageyears x 2.99) - (gender x 74.7). The value for gender is 0 in male subjects and 1 in female subjects.
Gait assessment: Stanmore questionnaire | 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  The Stanmore questionnaire has been used in the literature to assess functional outcome in patients with foot drop due to peroneal nerve injury. Seven sections (pain, need for orthosis, normal shoes, functional outcome, muscle power, degree of active dorsiflexion and foot posture) add up to a sum score of 100 points.
Gait assessment: Functional ambulation categories | 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  Functional ambulation categories (FAC) is a useful scale to assess gait in patients with foot drop. It is a six point scale, that is used in stroke literature and can help determine how much assistance a patient requires.
  FAC 0 reflects a nonfunctional state and FAC 5 equals a normal gait pattern.
Gait assessment: Gait speed as measured by the 10-meter walk test | 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  Walking speed is an important aspect of gait and is often used as an objective measure of functional mobility. The 10-meter walk test is a commonly used and validated tool to assess gait speed.
Health economic assessment: Work Productivity and Activity Impairment Questionnaire (WPAI) | 6 weeks and 6 months after randomization
  Health economic aspects of foot drop will be evaluated through the Work Productivity and Activity Impairment Questionnaire (WPAI). The WPAI is widely used and validated in multiple languages.
  The WPAI questionnaire consists of 6 questions with regard to professional activity during the past 7 days.
Complications and neurologic deficits: Surgical complications | 10 days, 6 weeks and 18 months after surgery
  A list of possible complications is made available to all participating centers. Unforeseen complications will be recorded as free-text.
Electrodiagnostics: evolution of conduction block at the level of the fibular head | 3 months and 9 months after randomization.
  All patients will have repeated electrodiagnostic examinations. The evolution of the conduction block at the level of the fibular head will be documented in the eCRF.
Patient-reported outcome measurements regarding health-related quality of life: 5 Level Euro Quality of Life 5 Dimensions (EQ5D-5L) | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  The EQ-5D 5L is a generic measure of health-related quality of life developed by the EuroQol Group. It is a validated measurement of quality of life widely used in different pathologies. The questionnaire is made up of two parts. The first part is descriptive and uses five different dimensions to score quality of life. These five dimensions are mobility, self-care, activities of the daily life, pain/discomfort and anxiety/depression. There are five different answer possibilities within each dimension, i.e. "no problem", "slight problem", "moderate problem", "severe problem" and "unable to". This renders 3125 different answer possibilities. The second part uses a visual analogue scale (VAS) to score the current health status of the patient, ranging from zero to one hundred. Zero corresponds to death and one hundred corresponds to a (subjective) perfect health status.
Health economic assessment: Return to work | 6 weeks
  Health economic aspects will also be evaluated through the assessment of return to work. We expect subgroups of patients with foot drop to be unable to work. Once the foot drop has improved (or fully recovered), we expect patients to be able to return to work and to not experience any more related problems (after their initial recovery). In this trial population foot drop does in general not represent a chronic condition with periods of relapse. Either the foot drop recovers enough to be able to work again, or the foot drop does not sufficiently recover to resume previous professional activities.
  Taking this into account, return to work seems to represent a very important measure. Patients will be asked about return to work at the study visit six weeks after randomization. To avoid recall bias, patients will be asked in advance to record the date of return to work. During baseline assessments, subjects will be questioned if they are incapacitated to work due to the foot drop and the
Gait assessment: The proportion of patients in both groups who reach minimal normal age- and sex-specific reference values for distance covered in meters during the six-minute walk test | 9 months after randomization
  The distance covered during the six-minute walk test (6MWT) is validated and clinically used in gait analysis.
  6MWT: patients are instructed to walk as far as possible within six minutes (strokes of 30 meters of more).
  The minimal age- and sex-specific normal 6MWD is defined as 82% of the applied reference equations for prediction of the 6MWD. The reference value that will be used is 6MWDpred(m) = 868.8 - (ageyears x 2.99) - (gender x 74.7). The value for gender is 0 in male subjects and 1 in female subjects.
Complications and neurologic deficits: Motor changes as assessed by the Medical Research Council Score (MRC-score) for ankle eversion | 10 days (surgery), 6 weeks, 3 months, 6 months, 9 months and 18 months (after randomization)
  Medical Research Council (MRC)-score as clinical assessment of muscle strength. MRC-score ranges from 0 to 5.
  0: no movement
  1. contraction of muscle, but no movement
  2. movement, but not against gravity
  3. movement against gravity, but not against resistance
  4. movement against resistance
  5. normal strength

CONTACTS AND LOCATIONS:
Overall Officials: Tom Theys, M.D.; Ph.D., Principal Investigator — Univeristy hospitals of Leuven
Locations (18):
- Belgium (17):
  - AZ Sint-Maarten, Mechelen, Antwerpen
  - AZ Turnhout, Turnhout, Antwerpen
  - Sint Augustinus, Wilrijk, Antwerpen
  - Jessa Ziekenhuis, Hasselt, Limburg
  - AZ Vesalius, Tongeren, Limburg
  - AZ Alma, Eeklo, Oost-Vlaanderen
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - AZ Groeninge, department of neurosurgery, Kortrijk, West-Vlaanderen
  - AZ Damiaan, Ostend, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen
  - Universitaire Ziekenhuizen Antwerpen, Antwerp
  - ULB Erasme, department of neurosurgery, Brussels
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, department of neurosurgery, Genk
  - University Hospitals Of Leuven, department of neurosurgery, Leuven
  - CHU de Liège, department of neurosurgery, Liège
- Leids Universitair Medisch Centrum, department of neurosurgery, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poage C, Roth C, Scott B. Peroneal Nerve Palsy: Evaluation and Management. J Am Acad Orthop Surg. 2016 Jan;24(1):1-10. doi: 10.5435/JAAOS-D-14-00420. PMID 26700629
- [Background] Broekx S, Weyns F. External neurolysis as a treatment for foot drop secondary to weight loss: a retrospective analysis of 200 cases. Acta Neurochir (Wien). 2018 Sep;160(9):1847-1856. doi: 10.1007/s00701-018-3614-9. Epub 2018 Jul 1. PMID 29961126
- [Background] Cruz-Martinez A, Arpa J, Palau F. Peroneal neuropathy after weight loss. J Peripher Nerv Syst. 2000 Jun;5(2):101-5. doi: 10.1046/j.1529-8027.2000.00007.x. PMID 10905469
- [Background] Khedr EM, Fawi G, Allah Abbas MA, El-Fetoh NA, Zaki AF, Gamea A. Prevalence of Common Types of Compression Neuropathies in Qena Governorate/Egypt: A Population-Based Survey. Neuroepidemiology. 2016;46(4):253-60. doi: 10.1159/000444641. Epub 2016 Mar 15. PMID 26974980
- [Background] Kandil MR, Darwish ES, Khedr EM, Sabry MM, Abdulah MA. A community-based epidemiological study of peripheral neuropathies in Assiut, Egypt. Neurol Res. 2012 Dec;34(10):960-6. doi: 10.1179/1743132812Y.0000000099. PMID 23146298
- [Background] Poppler LH, Bansal A, Groves A, Sacks G, Davidge K, Mackinnon SE. Abstract 65: Subclinical Peroneal Nerve Entrapment May be an Under-recognized Cause of Falls in Hospitalized Patients. Plast Reconstr Surg. 2014 Mar;133(3 Suppl):76. doi: 10.1097/01.prs.0000445098.29964.cf. No abstract available. PMID 25942176
- [Background] Aprile I, Caliandro P, La Torre G, Tonali P, Foschini M, Mondelli M, Bertolini C, Piazzini DB, Padua L. Multicenter study of peroneal mononeuropathy: clinical, neurophysiologic, and quality of life assessment. J Peripher Nerv Syst. 2005 Sep;10(3):259-68. doi: 10.1111/j.1085-9489.2005.10304.x. PMID 16221285
- [Background] Aprile I, Padua L, Padua R, D'Amico P, Meloni A, Caliandro P, Pauri F, Tonali P. Peroneal mononeuropathy: predisposing factors, and clinical and neurophysiological relationships. Neurol Sci. 2000 Dec;21(6):367-71. doi: 10.1007/s100720070052. PMID 11441574
- [Background] Aprile I, Tonali P, Caliandro P, Pazzaglia C, Foschini M, Di Stasio E, Mondelli M, Padua L; Italian CTS and other entrapments Study Group. Italian multicentre study of peroneal mononeuropathy: multiperspective follow-up. Neurol Sci. 2009 Feb;30(1):37-44. doi: 10.1007/s10072-009-0010-5. Epub 2009 Jan 20. PMID 19153647
- [Background] Aprile I, Caliandro P, Foschini M, Di Stasio E, Padua L; Italian CTS and other Entrapments Study Group; Mondelli M. Multicentre study of peroneal mononeuropathy: multiperspective follow-up of nonsurgical cases. J Peripher Nerv Syst. 2007 Sep;12(3):232-3. doi: 10.1111/j.1529-8027.2007.00145.x. No abstract available. PMID 17868251
- [Background] Berry H, Richardson PM. Common peroneal nerve palsy: a clinical and electrophysiological review. J Neurol Neurosurg Psychiatry. 1976 Dec;39(12):1162-71. doi: 10.1136/jnnp.39.12.1162. PMID 1011026
- [Background] Bsteh G, Wanschitz JV, Gruber H, Seppi K, Loscher WN. Prognosis and prognostic factors in non-traumatic acute-onset compressive mononeuropathies--radial and peroneal mononeuropathies. Eur J Neurol. 2013 Jun;20(6):981-5. doi: 10.1111/ene.12150. Epub 2013 Mar 26. PMID 23530751
- [Background] Sipahioglu S, Zehir S, Askar H, Isikan UE. Peroneal nerve palsy secondary to prolonged squatting in seasonal farmworkers. Acta Orthop Traumatol Turc. 2015;49(1):45-50. doi: 10.3944/AOTT.2015.14.0074. PMID 25803253
- [Background] Sangwan SS, Marya KM, Kundu ZS, Yadav V, Devgan A, Siwach RC. Compressive peroneal neuropathy during harvesting season in Indian farmers. Trop Doct. 2004 Oct;34(4):244-6. doi: 10.1177/004947550403400424. PMID 15510960
- [Background] Fares MY, Dimassi Z, Fares J, Musharrafieh U. Peroneal neuropathy and bariatric surgery: untying the knot. Int J Neurosci. 2020 Apr;130(4):417-423. doi: 10.1080/00207454.2019.1694926. Epub 2020 Jan 6. PMID 31735096
- [Background] Maalla R, Youssef M, Ben Lassoued N, Sebai MA, Essadam H. Peroneal nerve entrapment at the fibular head: outcomes of neurolysis. Orthop Traumatol Surg Res. 2013 Oct;99(6):719-22. doi: 10.1016/j.otsr.2013.05.004. Epub 2013 Aug 27. PMID 23988424
- [Background] Humphreys DB, Novak CB, Mackinnon SE. Patient outcome after common peroneal nerve decompression. J Neurosurg. 2007 Aug;107(2):314-8. doi: 10.3171/JNS-07/08/0314. PMID 17695385
- [Background] Kim DH, Murovic JA, Tiel RL, Kline DG. Management and outcomes in 318 operative common peroneal nerve lesions at the Louisiana State University Health Sciences Center. Neurosurgery. 2004 Jun;54(6):1421-8; discussion 1428-9. doi: 10.1227/01.neu.0000124752.40412.03. PMID 15157299
- [Background] Mitra A, Stern JD, Perrotta VJ, Moyer RA. Peroneal nerve entrapment in athletes. Ann Plast Surg. 1995 Oct;35(4):366-8. doi: 10.1097/00000637-199510000-00006. PMID 8585678
- [Background] Mont MA, Dellon AL, Chen F, Hungerford MW, Krackow KA, Hungerford DS. The operative treatment of peroneal nerve palsy. J Bone Joint Surg Am. 1996 Jun;78(6):863-9. PMID 8666604
- [Background] Morimoto D, Isu T, Kim K, Sugawara A, Yamazaki K, Chiba Y, Iwamoto N, Isobe M, Morita A. Microsurgical Decompression for Peroneal Nerve Entrapment Neuropathy. Neurol Med Chir (Tokyo). 2015;55(8):669-73. doi: 10.2176/nmc.oa.2014-0454. Epub 2015 Jul 31. PMID 26227056
- [Background] Ramanan M, Chandran KN. Common peroneal nerve decompression. ANZ J Surg. 2011 Oct;81(10):707-12. doi: 10.1111/j.1445-2197.2010.05607.x. PMID 22295311
- [Background] Tarabay B, Abdallah Y, Kobaiter-Maarrawi S, Yammine P, Maarrawi J. Outcome and Prognosis of Microsurgical Decompression in Idiopathic Severe Common Fibular Nerve Entrapment: Prospective Clinical Study. World Neurosurg. 2019 Jun;126:e281-e287. doi: 10.1016/j.wneu.2019.02.042. Epub 2019 Feb 26. PMID 30822592
- [Background] Nirenberg MS. A simple test to assist with the diagnosis of common fibular nerve entrapment and predict outcomes of surgical decompression. Acta Neurochir (Wien). 2020 Jun;162(6):1439-1444. doi: 10.1007/s00701-020-04344-3. Epub 2020 Apr 23. PMID 32328792
- [Background] Lale A, Kirkil C, Ozturk S, Yur M, Can OF, Artas G, Aygen E. The results of surgical decompression in the treatment of foot drop due to peroneal nerve entrapment after bariatric surgery. Surg Obes Relat Dis. 2020 Nov;16(11):1684-1691. doi: 10.1016/j.soard.2020.06.054. Epub 2020 Jul 15. PMID 32800521
- [Background] Wilson C, Yaacoub AP, Bakare A, Bo N, Aasar A, Barbaro NM. Peroneal nerve decompression: institutional review and meta-analysis to identify prognostic associations with favorable and unfavorable surgical outcomes. J Neurosurg Spine. 2019 Feb 8;30(5):714-721. doi: 10.3171/2018.10.SPINE18626. Print 2019 May 1. PMID 30738397
- [Background] Troosters T, Gosselink R, Decramer M. Six minute walking distance in healthy elderly subjects. Eur Respir J. 1999 Aug;14(2):270-4. doi: 10.1034/j.1399-3003.1999.14b06.x. PMID 10515400
- [Background] Gibbons WJ, Fruchter N, Sloan S, Levy RD. Reference values for a multiple repetition 6-minute walk test in healthy adults older than 20 years. J Cardiopulm Rehabil. 2001 Mar-Apr;21(2):87-93. doi: 10.1097/00008483-200103000-00005. PMID 11314289
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Derived] Oosterbos C, Rummens S, Bogaerts K, Van Hoylandt A, Hoornaert S, Weyns F, Dubuisson A, Ceuppens J, Schuind S, Groen JL, Lemmens R, Theys T. A randomized controlled trial comparing conservative versus surgical treatment in patients with foot drop due to peroneal nerve entrapment: results of an internal feasibility pilot study. Pilot Feasibility Stud. 2023 Oct 31;9(1):181. doi: 10.1186/s40814-023-01407-x. PMID 37908016
- [Derived] Oosterbos C, Rummens S, Bogaerts K, Hoornaert S, Weyns F, Dubuisson A, Lemmens R, Theys T. Conservative versus surgical treatment of foot drop in peroneal nerve entrapment: rationale and design of a prospective, multi-centre, randomized parallel-group controlled trial. Trials. 2022 Dec 30;23(1):1065. doi: 10.1186/s13063-022-07009-x. PMID 36581937

DOCUMENTS (1):
  • Study Protocol (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04695834/Prot_000.pdf